CLINICAL TRIAL: NCT03403608
Title: Subcutaneous Suppressive Antibiotic Therapy for Bone and Joint Infections
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: SSA therapy for BJI
Record Dates: First submitted 2017-11-20; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-11

CONDITIONS: Bone Infection; Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For patients having a bone or joint infections, with or without device, optimal surgical therapy could be sometimes non-feasible, especially in the elderly population. Therefore, a medical therapy with oral prolonged suppressive antibiotic therapy (PSAT) seems to be an option to prevent recurrence and prosthesis loosening.

Subcutaneous (SC) administration of injectable intravenous antibiotics as prolonged suppressive antibiotic therapy could be a convenient way when oral treatment is not available to facilitate ambulatory care, this practice being considered as routine care.

The aim of this study is to evaluate tolerance and efficacy of subcutaneous administration of antibiotics for prolonged suppressive antibiotic therapy in patients having this treatment as part of their routine care.

ELIGIBILITY:
Inclusion Criteria:

* patients having bone or joint infection,
* patients with or without device treated by sub-cutaneous prolonged antibiotic therapy

Exclusion Criteria:

* diabetic foot osteomyelitis
* pressure ulcer-associated osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having bone or joint infection, with or without device
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Description of sub-cutaneous administration of antibiotics for PSAT | 60 months
  In case of PSAT (prolonged suppressive antibiotic therapy), the duration could be several years.
  The data collected are: name of molecule, rough, posology, duration.

SECONDARY OUTCOMES:
Tolerance of sub-cutaneous administration of antibiotics for PSAT | 60 months
  In case of PSAT (prolonged suppressive antibiotic therapy), the duration could be several years.
  This outcome will focus on severe adverse events induced by this sub-cutaneous and prolonged antibiotic therapy.
  Qualification of an adverse event is made using the CTCAE terminology: this terminology attributes a grade for every adverse event. There are 5 grades and a grade refers to the severity of the adverse event. A severe adverse event has a grade >=3.
Efficacy of sub-cutaneous administration of antibiotics for PSAT | 60 months
  A treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence des Infections Ostéo-Articulaires complexes (CRIOAc Lyon), Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pouderoux C, Becker A, Goutelle S, Lustig S, Triffault-Fillit C, Daoud F, Fessy MH, Cohen S, Laurent F, Chidiac C, Valour F, Ferry T; Lyon Bone and Joint Infection Study Group. Subcutaneous suppressive antibiotic therapy for bone and joint infections: safety and outcome in a cohort of 10 patients. J Antimicrob Chemother. 2019 Jul 1;74(7):2060-2064. doi: 10.1093/jac/dkz104. PMID 31220276